CLINICAL TRIAL: NCT02028195
Title: The CORE-trial: a Pragmatic Randomized Controlled Trial in Primary Care Investigating Effectiveness and Cost-effectiveness of the Check Your Health Preventive Programme Offered Population-wide to 30-49 Years
Brief Title: Effectiveness and Cost-effectiveness of the Check Your Health Preventive Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Collaborators: Tryg Danmark (Unknown); Randers Municipality, Denmark (Other); Region MidtJylland Denmark (Other)
Responsible Party: Principal Investigator, Annelli Sandbæk, Professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tryg 7-11-0500
Record Dates: First submitted 2013-12-13; First posted 2014-01-07 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Health Promotion; Cardiovascular Disease; Physical Inactivity; Selfreported Quality of Health; Mental Health
Keywords: Health check; Health promotion; prevention diabetes; prevention cardiovascular disease; mental health
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health check (Experimental): The intervention consists of invitation for a behavioural and clinical examination followed by either (I) referral to a health promoting consultation in general practice (II) targeted behavioural programmes at the local Health Centre or (III ) no need for follow-up.
  Interventions: Other: Health check
- No invitation (No Intervention): The persons randomised to the control arm does not get invitation to a health care examination before time for follow up in the intervention group.

INTERVENTIONS:
Other: Health check — The program includes four components:
  Invitation: All participants receive invitation by mail and a prefixed appointment time. A web-based questionnaire including self-reported health (SF12), physical activity, smoking habits and alcohol use/behaviour has to be answered before Health Examination (HE).
  The HE include: Blood pressure, waist, weight, lung function test, lipid profile, HbA1c and fitness (Aastrand).
  Health profile pamphlet: The participant receives a pamphlet with the results. The persons are stratified into three groups (I) referral to a consultation in general practice (GP) (II) targeted behavioural programs at the health centre (HC) or (III ) no identified need for health promoting follow-up.
  Follow-up according to risk-profile: If referred to GP treatment of risk conditions or diseases will follow national guidelines. The GPs were paid 50 Euros per health interview.
  Arms: Health check

SUMMARY:
Check your health is a prevention intervention designed to create awareness and action on health condition with focus at physical activity at a population-level to 30-49 years of age. It consists of a behavioural and clinical examination followed by either (I) referral to a health promoting consultation in general practice (II) targeted behavioural programmes at the local Health Centre or (III ) no need for follow-up; stratified after risk-profile. The CORE trial (Check your health) aim to investigate effectiveness on health and social outcomes of the preventive health check and to establish the cost-effectiveness according to life years gained; direct costs and total health costs. A pragmatic cluster randomised controlled trial has been established to meet the aims and in total 10.600 individuals from 35 practices have been randomized in to two groups that will be invited in 2013-14 and 2017-18 respectively. The group offered the preventive health check in 2013-14 will constitute the intervention group and the group examined in 2017 - 18 the control group. A follow up of the intervention group in 2017 - 18 will provide data for the intention to treat analysis revealing the effect. Outcome measures are level of physical activity, risk of getting cardiovascular disease, sick leave and labor market attachment.

ELIGIBILITY:
Inclusion Criteria:

* all citizens living in Randers Municipality aged 30-49 on 1 January 2012, identified in the Danish Civil Registers (DCR) and randomised for health check in 2013 or 2017.

Exclusion Criteria:

* Terminal illness, reported by their GP is exclusion criteria for receiving invitation.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11000 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 4 years
  Physical activity level will be measured by 1) self-reported physical activity (days/week with minimum 30 minutes moderate physical activity) and 2) physical fitness, measured by Aastrands submaximal bike-test.
Modelled cardiovascular risk | 4 years
  Cardiovascular risk will be measured as a modelled risk of developing cardiovascular disease within 10 years and includes information on age, gender, smoking status, systolic blood pressure and total cholesterol.
Health related quality of life | 4 years
  Health related quality of life measured by The Medical Outcome Study Short Form 12 Health Survey (SF12)
Functional capacity | 4 years
  Functional capacity will be measured as affiliation to the labor market (work participation in the last year)and sick leave > 3 weeks.

OTHER OUTCOMES:
Health economy assessment | 4 years
  The economic benefits of the interventions will be assessed by comparing mean direct and total costs (direct and productivity costs), and expected life years gained (LYG) in the intervention group with the control group (within a period of four.

CONTACTS AND LOCATIONS:
Overall Officials: Annelli Sandbæk, Professor, Principal Investigator — University of Aarhus; Helle T Maindal, Professor, Principal Investigator — University of Aarhus
Locations (1):
- Department of Public Health, Aarhus, Denmark

REFERENCES:
- [Derived] Bjerregaard AL, Dalsgaard EM, Bruun NH, Norman K, Witte DR, Stovring H, Maindal HT, Sandbaek A. Effectiveness of the population-based 'check your health preventive programme' conducted in a primary care setting: a pragmatic randomised controlled trial. J Epidemiol Community Health. 2022 Jan;76(1):24-31. doi: 10.1136/jech-2021-216581. Epub 2021 Jun 18. PMID 34145078
- [Derived] Geyti C, Christensen KS, Dalsgaard EM, Bech BH, Gunn J, Maindal HT, Sandbaek A. Factors associated with non-initiation of mental healthcare after detection of poor mental health at a scheduled health check: a cohort study. BMJ Open. 2020 Oct 16;10(10):e037731. doi: 10.1136/bmjopen-2020-037731. PMID 33067280
- [Derived] Geyti C, Dalsgaard EM, Sandbaek A, Maindal HT, Christensen KS. Initiation and cessation of mental healthcare after mental health screening in primary care: a prospective cohort study. BMC Fam Pract. 2018 Nov 17;19(1):176. doi: 10.1186/s12875-018-0864-9. PMID 30447688
- [Derived] Maindal HT, Stovring H, Sandbaek A. Effectiveness of the population-based Check your health preventive programme conducted in primary care with 4 years follow-up [the CORE trial]: study protocol for a randomised controlled trial. Trials. 2014 Aug 29;15:341. doi: 10.1186/1745-6215-15-341. PMID 25169211

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT02028195/SAP_001.pdf